CLINICAL TRIAL: NCT00068913
Title: Investigation of Clinical Syndromes Associated With mtDNA Point Mutations: MELAS/DCA Clinical Trial
Brief Title: Evaluating the Effectiveness of a Dichloroacetate in MELAS Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P01HD032062 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: MELAS Syndrome
Keywords: Lactic Acidosis; Mitochondrial Disorder; Stroke; Seizure
MeSH Terms: conditions — MELAS Syndrome; Acidosis, Lactic; Mitochondrial Diseases; Stroke; Seizures | interventions — Dichloroacetic Acid

INTERVENTIONS:
Drug: Dichloroacetate

SUMMARY:
Patients with the MELAS syndrome experience devastating mental impairment. This study will evaluate the effectiveness of the drug dichloroacetate (DCA) to reduce the symptoms of MELAS.

DETAILED DESCRIPTION:
Although many organ systems are affected by mitochondrial (mt) DNA point mutations, the nervous system is particularly vulnerable. Maternally inherited mtDNA point mutations may cause chronic progressive encephalopathies and mental retardation. Patients with MELAS (mitochondrial myopathy, encephalopathy, lactic acidosis, and stroke-like episodes) syndrome have the A3243G point mutation and elevated brain lactate levels. Research has shown that lactic acidosis is associated with progressive impairment in patients with MELAS. This study will evaluate the effectiveness of DCA in lowering lactate levels and slowing the progression of MELAS.

Patients with the A3243G mitochondrial mutation and who have had either a stroke or a seizure will be enrolled in this study. Patients will be randomized to receive either DCA or a placebo. At a predetermined time point, patients receiving DCA will be switched to placebo and patients receiving placebo will be switched to DCA. Patients will have study visits every 3 months for 3 years. Study visits will include neurological exams, cognitive testing, nerve conduction tests, and MRIs. Study medicine, testing, hospitalization for research purposes, and travel expenses will be fully covered by the study.

ELIGIBILITY:
Inclusion Criteria

* A3243G mtDNA point mutation or maternally related to someone who has the mutation
* Symptomatic with MELAS, including previous seizure or stroke
* Certain laboratory values
* Ability to comply with the study protocol

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C De Vivo, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States